CLINICAL TRIAL: NCT06965595
Title: The Effect of Different Physiotherapy Methods Applied After Gynecological Abdominal Surgery on Postoperative Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Turkan Akbayrak, Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/012/013
Record Dates: First submitted 2025-03-28; First posted 2025-05-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gynecologic Surgeries; Physical Therapy; Women Health
Keywords: Gynecological abdominal surgery; postoperative routine care; physiotherapy and rehabilitation; vagal stimulation
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Routine Care (Experimental): This group will be the control group. Routine care practices carried out in the hospital (vital sign monitoring, administration of analgesics, anti-inflammatory and antibiotics when necessary, and mobilization starting from the 6th hour) will be applied and the data will be recorded.
  Interventions: Other: Routine care
- Rutin care + Physiotherapy (Active Comparator): In addition to routine care practices, this group will receive physiotherapy and rehabilitation. During the postoperative period, the intervention will be applied twice a day.
  Interventions: Other: Routine care + Physiotherapy
- Routine care + vagal stimulation (Active Comparator): In addition to routine care practices, this group will receive vagal stimulation. The stimulation will be applied to the cervical region at 10 Hz, 200 μs for 20 minutes, twice a day.
  Interventions: Other: Routine care + Vagal stimulation
- Routine care + Physiotherapy + Vagal stimulation (Active Comparator): In addition to routine care practices, this group will receive physiotherapy and rehabilitation, along with vagal stimulation.
  Interventions: Other: Routine care + Physiotherapy + Vagal stimulation

INTERVENTIONS:
Other: Routine care — This group will be the control group. Routine care practices carried out in the hospital (vital sign monitoring, administration of analgesics, anti-inflammatory and antibiotics when necessary, and mobilization starting from the 6th hour) will be applied and the data will be recorded.
  Arms: Routine Care
Other: Routine care + Physiotherapy — In addition to routine care practices, this group will receive physiotherapy and rehabilitation. During the postoperative period, the intervention will be applied twice a day.
  Posture training: Information about posture will be provided in different positions and training will be conducted.
  Breathing training (Diaphragmatic breathing, thoracic expansion exercises)
  In-bed mobilization (Lower and upper extremity exercises, foot-ankle exercises (dorsiflexion-plantar flexion / inversion-eversion), hip and knee flexion-extension exercises, cervical region joint range of motion and stretching exercises, upper extremity exercises (shoulder elevation, circumduction, elbow and wrist flexion-extension exercises), pelvic floor training and exercises)
  Out-of-bed mobilization (Sitting, standing, walking training after the 6th hour)
  Arms: Rutin care + Physiotherapy
Other: Routine care + Vagal stimulation — In addition to routine care practices, this group will receive vagal stimulation. The stimulation will be applied to the cervical region at 10 Hz, 200 μs for 20 minutes, twice a day.
  Arms: Routine care + vagal stimulation
Other: Routine care + Physiotherapy + Vagal stimulation — In addition to routine care practices, this group will receive physiotherapy and rehabilitation, along with vagal stimulation.
  Arms: Routine care + Physiotherapy + Vagal stimulation

SUMMARY:
Gynecological pelvic surgeries include procedures such as myomectomy, hysterectomy, and removal of ovarian cysts performed in the pelvic region of women. In the postoperative period following these surgeries, symptoms such as pain, decreased bowel motility, gastrointestinal problems, nausea, and vomiting are commonly observed. Effective management of these symptoms is important to accelerate the recovery process and improve the quality of life of patients.

This study is planned to evaluate the effectiveness of physiotherapy during the hospitalization period after gynecological abdominal surgery and to examine the effects of different approaches on postoperative symptoms.

In our study, participants who undergo gynecological abdominal surgery and meet the inclusion and exclusion criteria will be divided into four groups for intervention. In addition to routine care, interventions including physiotherapy, vagal stimulation, and a combination of physiotherapy and vagal stimulation will be applied from the postoperative period until discharge. The effects of these interventions on pain, bowel function, autonomic functions, pelvic floor function, and walking will be examined.

DETAILED DESCRIPTION:
Gynecological pelvic surgeries refer to procedures performed in the pelvic region of women. These surgeries include procedures such as myomectomy, hysterectomy, and the removal of ovarian cysts. Surgical procedures can be performed through abdominal or vaginal routes.

Various complications may occur during or after surgical operations . In the postoperative period, complaints such as pain, decreased bowel motility (e.g., paralytic ileus) , gastrointestinal problems, nausea and vomiting, and pneumonia may occur . At the same time, the occurrence of these complaints may also lead to a decrease in the patient's level of mobility .

There are different treatment approaches for symptoms that occur in the postoperative period. In particular, pain is among the primary complaints of patients. This acute pain may lead to chronic pain and the analgesic agents used may cause side effects such as sedation, nausea, and ileus .

Physiotherapy and rehabilitation practices for gastrointestinal problems and pain in the postoperative period include applications such as breathing exercises, mobilization, and connective tissue massage .

In a study by Zia and colleagues on the effectiveness of early physiotherapy applications, cases who underwent abdominal hysterectomy were divided into two groups as control and experimental. The experimental group received a comprehensive physiotherapy rehabilitation plan including patient education, breathing exercises, early mobilization, connective tissue manipulation, and transcutaneous electrical nerve stimulation (TENS), while the control group only performed walking (ambulation). It was shown that participants in the experimental group had a faster time to first gas passage and a higher rate of defecation within the first 3 days compared to the control group. As a result of the study, it is stated that early postoperative intervention has the potential to accelerate the recovery process .

In another study, the effect of kinesio taping and breathing exercises on pain in cases undergoing gynecological abdominal surgery was examined. The researchers divided the participants into four groups: kinesio taping, breathing exercises, kinesio taping with breathing exercises, and control group, and conducted interventions for 3 days postoperatively. Time to gas passage and defecation times were evaluated, and kinesio taping was found to be the group with the best improvement in pain and the earliest gas passage time. The group that received kinesio taping and breathing exercises also showed shorter gas passage times. As a result, kinesio taping and kinesio taping with breathing exercises can be used as non-invasive methods in the postoperative period .

Recently, the vagal stimulation technique has come to the forefront among applications for pain relief . This method has also been used in individuals with complaints of constipation . Stimulation of the vagus nerve can be provided through invasive and non-invasive methods.

In a study conducted by Shi and colleagues in 2021, 42 patients with constipation-predominant irritable bowel syndrome were divided into two groups and received auricular vagal stimulation and sham vagal stimulation treatments. In this study, which examined constipation and abdominal pain, positive results such as increased bowel motility and reduced pain were obtained after 4 weeks .

In another study involving patients with chronic low back pain, 60 patients were divided into two groups to receive either conventional rehabilitation and home exercises or transcutaneous auricular vagal nerve stimulation and home exercises. At the end of the 3-week treatment program, intra-group evaluation results showed positive effects on mobility, functional status, depression, and sleep in all groups .

This study is planned to evaluate the effectiveness of physiotherapy during the hospitalization period after gynecological abdominal surgery and to examine the effects of different approaches on postoperative symptoms.

ELIGIBILITY:
Inclusion Criteria

* Being 18 years of age or older
* Having undergone surgery due to a gynecological condition
* Having undergone one of the following operations: hysterectomy, hysterectomy + oophorectomy, or hysterectomy + salpingo-oophorectomy
* Having undergone abdominal surgery

Exclusion Criteria

* Development of any complications during or after surgery
* Presence of active malignancy
* Presence of severe organ failure
* Presence of uncontrolled cardiac or other systemic disorders
* Presence of neurological or cognitive diseases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain (VAS) | Day 1 and Day 2
  Pain will be assessed before and after each session. Visual Analog Scale (VAS) will be used for this. Minimum value is 0 and max value is 10. Ten is a higher pain. Zero means no pain.
Pain threshold measurement | Baseline and Day 2
  A digital algometer device will be used to determine the pain threshold.
Assessment of Autonomic Functions | Day 1 and Day 2
  The recording will be made with an ECG device.R-R waves will be examined.
Assessment of Autonomic Functions | Day 1 and Day 2
  heart rate collected before and after the session.
Assessment of Autonomic Functions | Day 1 and Day 2
  Blood Pressure collected before and after the session.
Assessment of Autonomic Functions | Day 1 and Day 2
  respiratory rate collected before and after the session.
Assessment of saturation (SpO₂) | Day 1 and Day 2
  arterial oxygen saturation (SpO₂) levels of participants will be evaluated. The unit of measurement will be the percentage of oxygen saturation.
Postoperative period | From enrollment to the end of treatment at 2 day
  The time when the first feeling of needing to pass gas time and defecation occurs will be noted.
The walking time | Postoperative
  The time of first walking will be noted.
First food intake | Postoperative
  The time of First food intake will be noted.
Take a medicine | Day 1 and Day 2
  Analgesics and other medications taken will be noted.
Umblikus | Day 1 and Day 2
  Umbilicus circumference will be measured with a tape measure.
xiphoid - pubis distance | day 1 and day 2
  The distance between the xiphoid and pubis will be measured with a tape measure. It will be noted in cm.
Postoperative period | Postoperative
  The time when the first feeling of needing to urinate occurs and the time when the feeling of micturition occurs will be noted.

SECONDARY OUTCOMES:
DETAILED STORIES OF THE PATIENTS | Before treatment
  Participants' age, height, weight, number and status of pregnancies (gravida, abortus, dilation & curettage, parity, number of living children, etc.), previous surgeries, medications used, comorbidities, chronic diseases, marital status, and current type of surgery will be assessed.
  Medical history, personal and family medical background, BMI, smoking habits, other lifestyle habits, and allergy status will also be evaluated.
Two minutes walk | Day 1 and Day 2
  The distance she can walk in two minutes will be recorded
Pelvic Floor | Day 1 and Day 2
  To assess the condition of the pelvic floor, researchers will evaluate it using the Visual Analog Scale (VAS). This assessment will address whether the participant can feel the pelvic region, as well as the presence of pain, discomfort, or incontinence. Min value is 0 . It means no sense and max value is 10. It means high score for question.
Pelvic Floor Distress Inventory-20 (PFDI-20) | Day1 and Day 2
  Pelvic floor symptoms will be evaluated using the Pelvic Floor Distress Inventory-20 (PFDI-20), which includes a separate subheading for these symptoms.The higher the score obtained from this questionnaire, the greater the degree of complaints about pelvic floor dysfunction.
Quality of Recovery-40 | Day 1 and Day 2
  It will be used to examine the recovery characteristics of the participants throughout the treatment process.Higher scores indicating higher levels of functioning or well-being.
Respiratory Function Test | Day 1 and Day 2
  It will be used to assess the patient's respiratory capacity.
Patient Satisfaction | Day 2
  Their satisfaction with the treatment will be evaluated.Minimum value is 0 and max value is 10. Ten is a higher satisfaction. Zero means no satisfaction.
Mini Mental Test | Before treatment
  It will be used to evaluate the cognitive status item included in the exclusion criteria.
Operation process | Baseline
  Information regarding the surgery (duration and time) will be noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan Unıversıty, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No